CLINICAL TRIAL: NCT07082296
Title: Use of an Internet-Based Cognitive Behavioral Therapy Platform to Carry Out an Intervention Aimed at Promoting Emotional Well-Being in the University and Research Community
Brief Title: iCBT to Promote Emotional Well-being in University and Research Communities: Feasibility and Acceptability Study
Acronym: iCBT-Academia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joaquim Radua (Other)
Responsible Party: Sponsor-Investigator, Joaquim Radua, Leader of the IMARD group, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Organization: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023BENES003
Record Dates: First submitted 2025-07-04; First posted 2025-07-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Emotional Well-being
Keywords: iCBT; subjective well-being; emotional well-being; anxiety; depression; feasibility; acceptability; academia; university and research community
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- University and Research Community (Experimental): Participants will receive the self-guided 4-week iCBT intervention.
  Interventions: Behavioral: iCBT-Academia

INTERVENTIONS:
Behavioral: iCBT-Academia — iCBT-Academia is a brief, self-guided, internet-based cognitive behavioral therapy (iCBT) program specifically tailored to address the real-life challenges faced by the university and research community. It consists of four modules, each designed to be completed over a week.

SUMMARY:
This study will evaluate a brief internet-based cognitive behavioral therapy (iCBT) program developed specifically for university students, researchers, and academic staff.

People in academic settings often face high levels of pressure and may experience psychological difficulties such as anxiety or excessive worry. However, access to psychological support adapted to the academic context is frequently limited.

This study investigates whether a short, self-guided online iCBT program can help promote emotional well-being in this population. The program is based on cognitive behavioral therapy principles and is designed to be completed in four weeks, with brief sessions four times per week that can be accessed on any device.

Participants will complete questionnaires before and after the intervention to assess the feasibility, acceptability, and safety of the program, as well as changes in emotional well-being.

The aim is to evaluate whether this digital intervention can serve as a useful, scalable tool to support emotional well-being in university and research environments.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility, acceptability, and potential effects of a brief, self-guided internet-based cognitive behavioral therapy (iCBT) program-iCBT-Academia-designed specifically for the university and research community. The intervention consists of four weekly modules delivered through a digital platform, with each module including short CBT-based lessons and practical exercises tailored to the academic context.

The study will use a single-group open-label design. Based on ICBT's previous open trials (see, for example, trials NCT03457714 or NCT03946098), 25 participants should be sufficient to estimate feasibility and preliminary effects. Participants will complete self-report questionnaires assessing various aspects of emotional well-being (positive and negative affect, life satisfaction, anxiety, and depression) before and after the intervention, as well as acceptability (TAAS) and potential adverse effects (NEQ) after the intervention. Retention, compliance, and participant feedback will also be evaluated.

This project seeks to explore whether such a digital intervention is a viable and scalable tool to support emotional well-being in academic environments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Ability to read in Catalan or Spanish.
* Undergraduate or master's student, PhD student, or teaching and researching staff.

Exclusion Criteria (for the primary analysis):

* Report that they are receiving psychological treatment or have a current mental disorder diagnosis.
* High subjective well-being and minimal symptoms of anxiety and depression at baseline, defined as scoring ≥20 on the Positive Affect subscale and <10 on the Negative Affect subscale of the International Positive and Negative Affect Schedule - Short Form (I-PANAS-SF), scoring ≥26 on the Satisfaction With Life Scale (SWLS), and scoring <5 on both the Generalized Anxiety Disorder 7-item scale (GAD-7) and the Patient Health Questionnaire-9 (PHQ-9).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
Retention/compliance rates | Post-intervention (4 weeks after commencing treatment)
  Retention/compliance rates refer to the proportion of participants who complete the study and follow the intervention as intended.
Acceptability | Post-intervention (4 weeks after commencing treatment)
  Acceptability will be measured using the Treatment Acceptability and Adherence Scale (TAAS), a brief self-report questionnaire that evaluates the acceptability of the psychological intervention from the participant's perspective. The TAAS consists of 10 items rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). To maintain comparability with the original scale, total scores (ranging from 10 to 50) will be linearly rescaled to range from 10 to 70. Higher scores indicate greater acceptability and adherence.

SECONDARY OUTCOMES:
Changes in affect | Pre-intervention and post-intervention (4 weeks after commencing treatment). In addition, the 4-item version will be administered at 1, 2, and 3 weeks after commencing treatment.
  Affect will be measured using the International Positive and Negative Affect Schedule - Short Form (I-PANAS-SF), a 10-item self-report questionnaire designed to assess positive and negative affect. It includes two subscales: Positive Affect and Negative Affect, each comprising 5 items. Participants rate each item on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). Subscale scores range from 5 to 25. Higher scores on the Positive Affect subscale indicate greater experience of positive emotions, while higher scores on the Negative Affect subscale indicate greater experience of negative emotions. An additional, shorter 4-item version, comprising items 6, 7, 8, and 9 (the two items with the highest factor loadings for positive affect and the two with the highest loadings for negative affect), will also be used.
Changes in life satisfaction | Pre-intervention and post-intervention (4 weeks after commencing treatment). In addition, the 2-item version will be administered at 1, 2, and 3 weeks after commencing treatment.
  Life satisfaction will be measured using the Satisfaction With Life Scale (SWLS), a brief self-report questionnaire that assesses the cognitive component of subjective well-being through participants' ratings of their overall life satisfaction. The SWLS consists of 5 items rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). To maintain comparability with the original scale, total scores (ranging from 5 to 25) will be linearly rescaled to range from 5 to 35. Higher scores indicate greater life satisfaction. An additional, shorter 2-item version comprising items 1 and 3 (the two items with the highest factor loadings), will also be used.
Changes in anxiety symptoms | Pre-intervention and post-intervention (4 weeks after commencing treatment). In addition, GAD-2 will be administered at 1, 2, and 3 weeks after commencing treatment.
  Anxiety symptoms will be measured using the Generalized Anxiety Disorder 7-item scale (GAD-7), a brief self-report questionnaire that assesses the severity of anxiety symptoms experienced over the past two weeks. Each of the 7 items is rated on a 4-point Likert scale (0 = not at all to 3 = nearly every day), with total scores ranging from 0 to 21. Higher scores indicate greater severity of anxiety symptoms. GAD-2, a shorter version with 2 items, will also be used.
Changes in depressive symptoms | Pre-intervention and post-intervention (4 weeks after commencing treatment). In addition, PHQ-2 will be administered at 1, 2, and 3 weeks after commencing treatment.
  Depressive symptoms will be measured using the Patient Health Questionnaire-9 (PHQ-9), a brief self-report questionnaire that assesses the severity of depressive symptoms over the past two weeks, based on DSM diagnostic criteria. Each of the 9 items is rated on a 4-point Likert scale (0 = not at all to 3 = nearly every day), with total scores ranging from 0 to 27. Higher scores indicate greater severity of depressive symptoms. PHQ-2, a shorter version with 2 items, will also be used.
Possible negative effects | Post-intervention (4 weeks after commencing treatment). In addition, the 5-item version will be administered at 1, 2, and 3 weeks after commencing treatment.
  Possible negative effects will be assessed using the Negative Effects Questionnaire (NEQ), a brief self-report instrument designed to evaluate negative effects experienced during or after a psychological intervention. The version used includes 20 items covering five domains: symptoms, quality, dependency, stigma, and hopelessness. Each item captures two dimensions: (1) whether the effect occurred and was attributed to the intervention, and (2) the perceived negative impact, rated on a 5-point Likert scale from 1 (not at all) to 5 (extremely). Total impact scores range from 20 to 100, with higher scores indicating greater perceived negative effects. In addition, a shorter 5-item version-comprising items 6, 11, 12, 14, and 16 (the items with the highest factor loading in each domain and retained in the NEQ-20)-will also be used.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Radua, Principal Investigator — Institut d'Investigacions Biomèdiques August Pi i Sunyer
Locations (1):
- IDIBAPS, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No